CLINICAL TRIAL: NCT02392273
Title: A Prospective Observational Registry of Primary Headache Patients Treated With Ausanil
Status: Terminated | Type: Observational
Why Stopped: Study unable to recruit
Sponsor: VR1 Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: Ausanil Study 001
Record Dates: First submitted 2015-03-12; First posted 2015-03-18 (Estimated); Last update posted 2016-12-28 (Estimated); Status verified 2016-12

CONDITIONS: Primary Headache Disorders
Keywords: migraine; cluster headache; primary headache; Ausanil; capsicum annuum
MeSH Terms: conditions — Headache Disorders, Primary; Migraine Disorders; Cluster Headache

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Ausanil — Patients with Primary Headache disorders will receive Ausanil in the context of usual and routine clinical care.
  Other Names: capsicum annuum

SUMMARY:
This study is an observational study with the primary objective to assess the safety and tolerability of Ausanil in the treatment of primary headache disorders. The secondary objective is to assess headache pain, functional outcome, time loss to headache and patient satisfaction with Ausanil treatment.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 to 80 years
* Primary Headache disorder as per International Classification of Headache Disorders-11
* Ausanil naive
* Signed dated informed consent
* Females of childbearing potential must be using adequate contraception during study period.
* Willing and able to comply with registry requirements to document headache response

Exclusion Criteria:

* Known allergy to Ausanil or any of its ingredients
* Active bronchial asthma that in the opinion of the investigator would interfere with use of Ausanil
* Nasal obstruction due to any cause or extensive nasal surgery resulting in scarring or other such impact on nasal mucosa that might lead to heightened sensitivity to Ausanil in the opinion of the investigator.
* Pregnant or breast feeding females
* History of addictive behavior
* Any severe or chronic unstable medical or psychiatric condition
* Active nasal infection or inflammation
* Unable or unwilling to provide informed consent
* Suffer from atypical, basilar or hemiplegic migraine that is new onset or unstable.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in a Clinical headache practice (outpatient) with a diagnosis of a primary headache disorder.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-02; Primary Completion 2016-12 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events (all cause) | 8 weeks
  Patient/Physician reporting
Incidence of Adverse Events causally related to Ausanil | 8 weeks
  Patient/Physician reporting
Serious Adverse Events | 8 weeks
  Patient/Physician reporting

SECONDARY OUTCOMES:
Headache Response to Ausanil | 24 hours
  Change in Headache severity on a four point scale (0-3) will be measured at 5 minutes, one hour, two hours and twenty four hours
Functional Assessment | 24 Hours
  Improvement in ability to function after Headache treatment
Patient satisfaction for Treatment | 24 hours
  Patients will be asked to rate their satisfaction with treatment on a 7 point scale (very dissatisfied to very satisfied)
Time Loss to headache | 24 hours
  How many hours of function were lost as result of the headache?
Use of Rescue Medication | 24 hours
  Frequency of Rescue medication will be tabulated
Sting severity and duration | one hour
  How long does the sting associated with Ausanil treatment last?

CONTACTS AND LOCATIONS:
Overall Officials: Seth Stoller, MD, Principal Investigator — Atlantic Health System
Locations (1):
- Atlantic Health System/Overlook Medical Center Medical Arts Center, Summit, New Jersey, United States